CLINICAL TRIAL: NCT03837795
Title: The Efficiency of Neurofeedback Therapy for Enhancing Participation in Occupations, Decreasing Pain Sensitivity, Improving Life Satisfaction and Brain Neural Activity in Adults With Sensory Over Responsivity - a Pilot Study
Brief Title: Examining the Efficiency of Neurofeedback Therapy on Adults With Sensory Over Responsivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Tami Bar-Shalita, Principal Investigator, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1710.18
Record Dates: First submitted 2019-01-08; First posted 2019-02-12 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sensory Modulation Disorder; Sensory Over-Responsivity
Keywords: Neurofeedback; Sensory Modulation Disorder; Sensory Over-Responsivity

STUDY DESIGN:
Intervention Model Description: it is a serial experimental research design, which includes 10 individuals with sensory over responsivity aged 21-45 years will participate
Masking Description: The researcher that will perform the measurement assessments will differ from the one that will provide the therapy sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback therapy group (Experimental)
  Interventions: Device: Neurofeedback treatment

INTERVENTIONS:
Device: Neurofeedback treatment — A treatment that developed to train adults with sensory modulation disorder by applying EEG (Curry 7 EEG system, Neuroscan-Compumedics). This treatment will aim to normalize the Alpha power (amplitude).

SUMMARY:
Sensory Over-Responsivity (SOR) is characterized by a disruption in regulating sensory stimuli and can significantly impact pain perception and restrict daily participation and quality of life. Altered neurophysiological processes in SOR are documented, revealing reduced electroencephalogram at rest and P300 amplitudes, the latter tested through event-related potentials (ERP). Both may explain the failure to regulate incoming sensory stimuli. Neurofeedback (NF) therapy, a remedial treatment approach, aims at self-regulating the brain's neural activity and has proven its efficiency in treating comorbid SMD syndromes.

Our study aims to investigate NF therapy efficiency in decreasing pain sensitivity, enhancing auditory ERP components of P300, increasing the power of the alpha band, life-satisfaction and Goal Attainment Scaling (GAS) scores in adults with SOR.

DETAILED DESCRIPTION:
In this serial experimental research design, 10 individuals with SOR aged 21-45 years will participate. A medical and demographic questionnaire and the Sensory Responsiveness Questionnaire-Intensity Scale (SRQ-IS) will be applied to screen for participation eligibility. Outcome measures will be conducted at 4-time points (1. baseline- 3 weeks pre-treatment; 2. before the first treatment session; 3. after the last treatment session; and 4. a month post-treatment) applying: The Goal Attainment Scaling (GAS), the P300 component using a neurophysiological assessment of the 'Oddball paradigm', the alpha power using electroencephalogram resting state, and electronic versions of the Satisfaction with Life Scale, the World Health Organization Disability Assessment Schedule, and the Pain Sensitivity Questionnaire. Sixteen individually therapy sessions of 45 minutes each, twice a week, will be held at the same time of day.

Repeated measures ANOVA or a non-parametric equivalent will be used to analyze the dependent variables measures change over time.

ELIGIBILITY:
Inclusion Criteria:

1. Having SOR indicated by a score higher than 2.39 on the Sensory Responsiveness Questionnaire-Aversive scale.
2. free of analgesic medicines for no less than 24 hours before the sessions.
3. independent functioning in the community.
4. fluency in understanding and reading Hebrew

Exclusion Criteria:

1. metabolic, psychiatric, neurological, or neuro-developmental, but ADHD diagnosis
2. acute or chronic pain.
3. regular intake of neurological, psychiatric and analgesic medicines.
4. participating in other therapies (i.e., cognitive therapies) at present.
5. substance abuse.
6. pregnancy.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
The Satisfaction with Life Scale (SWLS) | assesses the change between the baseline (3 weeks pre-treatment), and after 28 days from the last treatment session
  assesses global life satisfaction
Goal Attainment Scaling (GAS) | assesses the change between the baseline (3 weeks pre-treatment), and after 28 days from the last treatment session
  a standardized therapeutic method used to evaluate the participants' progress toward their functional goals
The World Health Organization Disability Assessment Schedule (WHODAS-2.0) | assesses the change between the baseline (3 weeks pre-treatment), and after 28 days from the last treatment session
  To evaluate participants' participation level in the last month

SECONDARY OUTCOMES:
Pain Sensitivity Questionnaire (PSQ) | 3 weeks pre-treatment, 2 days before first treatment session, two days after the last treatment session and after month of the treatment
  a standardized self-report questionnaire assessing daily pain sensitivity
Electroencephalogram (EEG) Resting State | 3 weeks pre-treatment, 2 days before first treatment session, two days after the last treatment session and after month of the treatment
  To measure alpha band (8-12Hz) power

OTHER OUTCOMES:
Auditory Evoked Related Potentials (AERP) | 3 weeks pre-treatment, 2 days before first treatment session, two days after the last treatment session and after month of the treatment
  Change from Baseline to 28 days after the last treatment session: An EEG method will be used to evaluate the brain responses to auditory stimulus.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Tami Bar-Shalita, Tel Aviv, Israel